CLINICAL TRIAL: NCT03063749
Title: A Post-approval Study of the Medtronic Resolute Onyx™ Zotarolimus-Eluting Coronary Stent System
Brief Title: RESOLUTE ONYX Post-Approval Study
Acronym: ONYX PAS
Status: Completed | Type: Observational
Sponsor: Medtronic Vascular (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT16025RES003
Record Dates: First submitted 2017-02-21; First posted 2017-02-24 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Primary Cohort: Subjects receiving stents 2.0 mm - 4.0 mm in diameter will be included in the Primary Cohort.
  Interventions: Device: Resolute Onyx™ Zotarolimus-Eluting Coronary Stent System
- Extra Large Vessel (XLV) Cohort.: Subjects receiving stents 4.5 mm or 5.0 mm in diameter will be included in the Extra Large Vessel (XLV) Cohort.
  Interventions: Device: Resolute Onyx™ Zotarolimus-Eluting Coronary Stent System

INTERVENTIONS:
Device: Resolute Onyx™ Zotarolimus-Eluting Coronary Stent System — Medtronic Resolute Onyx™ Zotarolimus-Eluting Coronary Stent System, sizes 2.0 mm - 4.0 mm
  Groups: Primary Cohort
Device: Resolute Onyx™ Zotarolimus-Eluting Coronary Stent System — Medtronic Resolute Onyx™ Zotarolimus-Eluting Coronary Stent System, sizes 4.5 mm - 5.0 mm
  Groups: Extra Large Vessel (XLV) Cohort.

SUMMARY:
To observe the continued performance of the Medtronic Resolute Onyx™ Zotarolimus-Eluting Coronary Stent System in a real-world more-comer population.

ELIGIBILITY:
Key Inclusion Criteria

* Symptomatic coronary artery disease including subjects with chronic stable angina, silent ischemia, and acute coronary syndromes including non-ST elevation and ST-elevation myocardial infarction
* Subject is an acceptable candidate for treatment with a drug eluting stent in accordance with the applicable guidelines on percutaneous coronary interventions, manufacturer's Instructions for Use, and the Declaration of Helsinki

Key Exclusion Criteria

* Unprotected left main disease
* Subjects with planned PCI of three vessel disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The device will be used in subjects meeting the inclusion and exclusion criteria according to the Instructions for Use.
Sampling Method: Non-Probability Sample
Enrollment: 416 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2018-10-20 (Actual); Study Completion 2022-08-18 (Actual)

PRIMARY OUTCOMES:
Target Lesion Failure | 12 months
  Target Lesion Failure (TLF), defined as cardiac death, target vessel myocardial infarction (Q wave and non-Q wave), or clinically driven target lesion revascularization (TLR) by percutaneous or surgical methods

SECONDARY OUTCOMES:
Acute Success (Device, Lesion, Procedure) | 30 days and 6, 12, 24, and 36 months post-procedure
  Acute Success (Device, Lesion, Procedure)
Cardiac Death | 30 days and 6, 12, 24, and 36 months post-procedure
  Cardiac Death
Target Vessel Myocardial Infarction (TVMI) | 30 days and 6, 12, 24, and 36 months post-procedure
  Target Vessel Myocardial Infarction (TVMI)
Target Lesion Revascularization (TLR) | 30 days and 6, 12, 24, and 36 months post-procedure
  Target Lesion Revascularization (TLR)
Target Vessel Revascularization (TVR) | 30 days and 6, 12, 24, and 36 months post-procedure
  Target Vessel Revascularization (TVR)
Cardiac Death and TVMI | 30 days and 6, 12, 24, and 36 months post-procedure
  Cardiac Death and TVMI
Major Adverse Cardiac Event (MACE) | 30 days and 6, 12, 24, and 36 months post-procedure
  Defined as death, myocardial infarction (Q wave and non-Q wave), emergent coronary bypass surgery, or clinically-driven repeat target lesion revascularization by percutaneous or surgical methods
Target Lesion Failure (TLF) | 30 days and 6, 12, 24, and 36 months post-procedure
  Target Lesion Failure (TLF)
Target Vessel Failure (TVF) | 30 days and 6, 12, 24, and 36 months post-procedure
  Target Vessel Failure (TVF)
Stent Thrombosis (ST) | 30 days and 6, 12, 24, and 36 months post-procedure
  Stent Thrombosis (ST)

CONTACTS AND LOCATIONS:
Locations (28):
- United States (23):
  - Huntsville Hospital, Huntsville, Alabama
  - Scripps Green Hospital, La Jolla, California
  - Riverside Community Hospital, Riverside, California
  - Hartford Hospital, Hartford, Connecticut
  - Morton Plant Hospital, Clearwater, Florida
  - North Florida Regional Medical Center, Gainesville, Florida
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - WellStar Kennestone Hospital, Marietta, Georgia
  - University of Michigan Health System - University Hospital, Ann Arbor, Michigan
  - Mercy Hospital (Coon Rapids MN), Coon Rapids, Minnesota
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Nebraska Medicine, Omaha, Nebraska
  - Desert Springs Hospital Medical Center, Las Vegas, Nevada
  - North Shore University Hospital, Manhasset, New York
  - NYU Langone Medical Center, New York, New York
  - Columbia University Medical Center/NewYork Presbyterian Hospital, New York, New York
  - Saint Joseph's Hospital Health Center, Syracuse, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Baptist Memorial Hospital-Memphis, Memphis, Tennessee
  - TriStar Centennial Medical Center, Nashville, Tennessee
  - Houston Methodist Hospital, Houston, Texas
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Saint Vincent Hospital (Green Bay WI), Green Bay, Wisconsin
- Belgium (2):
  - C.H.U. de Charleroi, Charleroi
  - Ziekenhuis Oost Limburg - Campus Sint-Jan, Genk
- France (2):
  - Centre Hospitalier Universitaire Besancon - Hôpital Jean Minjoz, Besançon
  - CHU Toulouse - Hôpital Rangueil, Toulouse
- Stredoslovensky Ustav Srdcovych a Cievnych Chorob a.s, Banská Bystrica, Slovakia